CLINICAL TRIAL: NCT05724030
Title: Effect of Integrated Pulmonary Index on Hypoxia
Brief Title: Use of Integrated Pulmonary Index Monitorisation in Children Undergoing Botulinum Toxin Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Zehra Ipek ARSLAN, Professor, Turkish Society of Anesthesiology and Reanimation
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: KAEK/26.bl.06
Record Dates: First submitted 2023-01-24; First posted 2023-02-13 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2023-12

CONDITIONS: Cerebral Palsy; Pediatric ALL
Keywords: botilinum toxin; pediatrics; ıntegrated pulmonary index; hypoxia
MeSH Terms: conditions — Cerebral Palsy; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Hypoxia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- integrated pulmonary index hypoxia -capnogarph (Active Comparator): integrated pulmonary index montorization apliied
  Interventions: Device: integrated pulmonary index; Device: saturation
- saturation - apnea (Experimental): saturation apllied
  Interventions: Device: integrated pulmonary index; Device: saturation

INTERVENTIONS:
Device: integrated pulmonary index — integarted pumobary index monitoring
Device: saturation — saturation monitorization

SUMMARY:
This study aimed to detect hypoxia early with ıntegrated pulmonary index monitoring compared to saturation.

DETAILED DESCRIPTION:
This trial will be held at the kocaeli Universty Hospital. 75 children 4-17 years of age undergoing botulinum toxin injection with sedation will be enrolled in this prospective study. Patients premedicated with midasolam iv 0.5 mg bolus and then sedated with propofol 1 mg/kg and fentanyl 0.5 mg/kg . Integrated pulmonary monitoring and noninvasive capnograhy will be used. Bis monitoring and spo2 monitoring will be applied. standard anesthesia monitoring including noninvasive blood pressure, spo2 , ekg and heart rate will be monitored. This trial aimed to detect hypoxia and apnea earlier than pulse oximetry.

ELIGIBILITY:
Inclusion Criteria:

* 4-16 age pediatrics
* undergoing botilinum injection with sedation
* asa 1-2

Exclusion Criteria:

* > 18 age
* asa 3-4
* patients with upper respiratory tract infection

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 69 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2024-09-03 (Actual); Study Completion 2024-10-11 (Actual)

PRIMARY OUTCOMES:
hypoxia | 20 seconds
  desaturation spo2 below 90

SECONDARY OUTCOMES:
apnea - ıntegrated pulmonary index | 20 seconds
  no respiration ıntegrated pulmonary index under 4

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University School of Medicine, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No